CLINICAL TRIAL: NCT02643836
Title: Pulsed Electromagnetic Field (PEMF) Therapy for Post-Concussive Syndrome
Acronym: PEMF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Rio Grande Neurosciences (Industry)
Responsible Party: Principal Investigator, Ross D. Zafonte, MD, Head of the Department of Physical Medicine and Rehabilitation, Harvard Medical School, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014D006902
Record Dates: First submitted 2015-10-08; First posted 2015-12-31 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Post Concussive Syndrome; Concussion
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment PEMF (Experimental): The investigators will recruit and enroll 76 patients (between 18 and 30 years of age) who have had persistent symptoms consistent with PCS for at least 4 weeks, but not more than 6 months, after the initial injury. The experimental group will contain 38 subjects. Each study subject will receive two hats, which contain the integrated PEMF device, this will be done to ensure continuity of treatment in case that one of the hats stops working due to the battery running out. The subjects will receive PEMF treatment for 15 minutes three times per day for 6 weeks. Upon enrollment and at the end of the 6-week treatment period, all subjects will undergo a comprehensive assessment that will include symptom inventories, neuropsychological tests, qEEG measurement and near-infrared spectroscopy. The investigators will conduct a 3-month follow-up to assess longer-term outcomes.
  Interventions: Device: PEMF
- Sham Treatment (Sham Comparator): The investigators will recruit and enroll 76 patients (between 18 and 30 years of age) who have had persistent symptoms consistent with PCS for at least 4 weeks, but not more than 6 months, after the initial injury. The sham group will contain 38 subjects. Each study subject will receive two hats, which contain a de-activated PEMF device, the device will still be blinking to show sham treatment activity. The sham subjects will receive the sham treatment for 15 minutes three times per day for 6 weeks. Upon enrollment and at the end of the 6-week treatment period, all subjects will undergo a comprehensive assessment that will include symptom inventories, neuropsychological tests, qEEG measurement and near-infrared spectroscopy. The investigators will conduct a 3-month follow-up to assess longer-term outcomes.
  Interventions: Device: PEMF

INTERVENTIONS:
Device: PEMF — The PEMF device (Rio Grande Neurosciences - RGN) the investigators would be testing has been shown to have significant anti-inflammatory effects in animals and humans and an excellent safety profile in several clinical studies. Key findings demonstrated that PEMF-treated rodents with a closed-head TBI exhibited a 5-fold decrease in IL-1b in the cerebral spinal fluid, an outcome associated with decreased neuropathology and improved function.
  Other Names: Pulsed Electromagnetic Field Therapy

SUMMARY:
The objectives are to evaluate impact of Pulsed electromagnetic field (PEMF) therapy on patients with Post-Concussive Syndrome with Rivermead Post Concussion Symptom Questionnaire (RPQ) as a primary outcome, followed by fatigue and mood as second and tertiary outcomes respectively. The investigators will also investigate brain tissue activity and oxygenation by evaluating brain wave activity via non-invasive quantitative electroencephalogram and near infrared spectroscopy testing pre and post study to better understand the metabolic effect of the PEMF intervention.

The investigators hypothesize that the PEMF treatment will have an effect on improvement of brain metabolism as measured by Near Infrared Spectroscopy which will in turn assist with improvement of the chronic symptoms of cognitive deficits, mood and fatigue as related to Post-Concussive Syndrome.

DETAILED DESCRIPTION:
76 subjects will be enrolled for this experiment. Each subject will go through the screening procedure as outlined above. After consent and screening are complete each subject will receive a hat that delivers three 15 minute stimulations per day for the duration of 6 weeks. Each study subject will receive two hats, which contain the integrated PEMF device, this will be done to ensure continuity of treatment in case that one of the hats stops working due to the battery running out.

The PEMF device to be used will be an investigational, battery powered custom-made stimulator able to deliver an electromagnetic field. This device operates at very low amplitude (0.05 gauss magnetic field strength) and requires only watch batteries for power, which allows the technology to be portable (e.g., used at home), versatile, inexpensive, and safe, (vi) we have integrated the PEMF device into a wearable baseball hat to improve tolerance and compliance and can also monitor patient use in this configuration.

The study device consists of a printed circuit board PEMF signal generator and an AAA battery-driven power supply encased in high density plastic, a solid wire-loop antenna covered in medical grade silicone, all of which are built into a standard baseball-style cap, with the antenna fitted around its largest internal circumference. The device was designed to be easily used and is activated by donning the cap. Once donned, a 15-minute treatment cycle starts and stops automatically. The device requires at least 2 hours between treatments, and cannot be activated again until that period has elapsed. A light on the power supply blinks while the unit is active. EEG and NIR will be obtained at visits 1, 2 and at three month follow up to better evaluate brain oxygenation and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* History of a mild or moderate traumatic brain injury in the previous 6 months related to a sports injury
* Symptomatic Rivermead Postconcussion Symptom Questionnaire (RPQ) scores (RPQ 3 > 3, RPQ 13 >8)
* Age 18-30
* Willing and able to sign informed consent
* Willing and able to attend all study assessments

Exclusion Criteria:

* Severe traumatic brain injury defined by a post-injury Glasgow Coma Scale score ≤ 8 greater than 30 minutes following the injury or post-traumatic amnesia lasting longer than 1 week
* Time since injury less than 4 weeks or greater than 6 months
* Any concussion that is not sustained during sports activity
* Concussions sustained during mixed martial arts or boxing activities
* Positive CT scan or MRI related to brain injury
* Recently beginning methylphenidate or amphetamine-dextroamphetamine treatment within two months
* Pre-existing diagnosis of learning disability or neurodevelopmental disorder (other than ADD/ADHD)
* Pre-existing significant neurological disorder (e.g., seizures, CNS neoplasms) or history of neurosurgical intervention
* Prior psychiatric hospitalization
* Current substance abuse or dependence (AUDIT-C)
* Pacemaker
* Implanted stimulation devices
* Pregnant
* Unstable medical conditions
* Unable to read and/or understand the purpose and participating conditions of the study
* Any condition that would prevent participation in study procedures or condition the investigator believes would make the subject unsuitable for participation in the study.
* Non-English speaking

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Rivermead Post-Concussion Symptom Questionnaire | 5 minutes
  basic post-concussion questionaire

SECONDARY OUTCOMES:
Ruff Neurobehavioral Inventory | 6 minutes
  basic neurobehavioral inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ross Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital

REFERENCES:
- [Result] Boake C, McCauley SR, Levin HS, Pedroza C, Contant CF, Song JX, Brown SA, Goodman H, Brundage SI, Diaz-Marchan PJ. Diagnostic criteria for postconcussional syndrome after mild to moderate traumatic brain injury. J Neuropsychiatry Clin Neurosci. 2005 Summer;17(3):350-6. doi: 10.1176/jnp.17.3.350. PMID 16179657